CLINICAL TRIAL: NCT04434976
Title: Delayed Diagnosis of Bacteriologically Positive Pulmonary Tuberculosis and Relative Optimized Suggestions in China
Status: Completed | Type: Observational
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, Wen-hong Zhang, Director of Division of Infectious Diseases, Huashan Hospital
Other Study IDs: KY-2019TB-20
Record Dates: First submitted 2020-06-14; First posted 2020-06-17 (Actual); Last update posted 2020-06-17 (Actual); Status verified 2020-06

CONDITIONS: Tuberculosis; Pulmonary, Confirmed, Unspecified Means
Keywords: bacteriologically confirmed pulmonary tuberculosis; health-seeking pathways; Delayed Diagnosis
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- delayed diagnosis: The length from the first clinical visit date to the diagnosis confirmed date is more than 14 days. Diagnosis is confirmed by any positive result of anti fast bacteria smear, culture, histological test, and molecular detection such as GeneXpert.
- undelayed diagnosis: The length from the first clinical visit date to the diagnosis confirmed date is equal or less than 14 days. Diagnosis is confirmed by any positive result of anti fast bacteria smear, culture, histological test, and molecular detection such as GeneXpert.

SUMMARY:
The purpose of the study is to collect health-seeking pathways, sociodemographic characteristics and symptoms of 400 newly diagnosed patients with bacteriologically confirmed pulmonary tuberculosis(TB).

DETAILED DESCRIPTION:
This research is a retrospective, multicenter, case-control study. The purpose of this study is to collect and assess health-seeking pathways, sociodemographic characteristics and symptoms of 400 newly diagnosed patients with bacteriologically confirmed pulmonary tuberculosis(TB).

According to inclusion criteria and exclusion criteria, a total of 400 participants with bacteriologically confirmed TB will be recruited and acquired their health-seeking pathways in different clinical institutions of pulmonary tuberculosis. Totally, 20 TB-designated medical institutions will be conducted in depth, covering the eastern region (7), the central region (8) and the western region (5), each hospital will enroll 20 eligible patients on the basis of convenience.

The cohorts are divided into delayed diagnosis and undelayed diagnosis. The former is defined if The length from the first clinical visit date to the diagnosis confirmed date is more than 14 days. Diagnosis is confirmed by any positive result of anti fast bacteria smear, culture, histological test, and molecular detection such as GeneXpert. By offline or online interview, we aim to collect basic sociodemographic characteristics, symptoms, health-seeking pathway, including: hospital name, the date of each visit, laboratory tests and radiology evaluation results, diagnosis, treatment, medical and transportation costs. Then list the hospitals of previous consultations and trace their classification through the official website of the Health and Medical Commission. Determine whether these hospital are designated institution based on the CDC's publicity. Consult the laboratory facilities by phone.

The primary objective is to gain the median time of pulmonary tuberculosis diagnosis confirmed and the correlation between the classification of the first-visit-institution and the diagnosis delay of the pulmonary tuberculosis.

The secondary objective is to gain the bacteriology examination coverage rate: anti fast bacteria smear, tuberculosis culture, and GeneXpert; the correlation between the use of fluoroquinolones as anti-infection treatment before tuberculosis diagnosis confirmed and the diagnosis delay of the pulmonary tuberculosis; the sociodemographic characteristics of patients with or without pulmonary tuberculosis diagnosis delay; The rates of onset symptoms and its correlation to diagnosis delayed of pulmonary tuberculosis diagnosis confirmed patients.

ELIGIBILITY:
Inclusion Criteria:

* Bacteriological positive: including positive AFB smear/ culture / molecular test;
* Agree to accept this survey;

Exclusion Criteria:

* HIV antibody positive and AIDS patients;
* Combined with extrapulmonary TB;
* Critically ill patients, and according to the judgment of the research physician, it is impossible to survive for more than 16 weeks;

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: In the study, 400 patients with bacteriologically confirmed pulmonary tuberculosis(TB) were chose from 20 hospitals, each hospital select 20 patients according to the eligibility criteria randomly. These 20 TB-designated medical institutions are covering the eastern region (7), the central region (8) and the western region (5) among China.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2019-09-08 (Actual); Primary Completion 2019-11-02 (Actual); Study Completion 2020-01-10 (Actual)

PRIMARY OUTCOMES:
The median time of pulmonary tuberculosis diagnosis confirmed | immediately after asking the medical history and collecting the result of TB diagnosis
  Time from the date of patients' symptoms onset to the date of pulmonary tuberculosis diagnosis confirmed
The correlation between the classification of the first-visit-institution and the diagnosis delay of the pulmonary tuberculosis | immediately after asking the medical history and collecting the result of TB diagnosis
  We collect the classification and the quality of the first-visit-institution of diagnosis confirmed patients by asking the past medical histories. According to the evidence of duration from symptoms onset to pulmonary TB diagnosis confirmed, use logistic correlation to find the relation between the classification of the first-visit-institution and the diagnosis delay.

SECONDARY OUTCOMES:
Bacteriology examination coverage rate: anti fast bacteria smear, tuberculosis culture, and GeneXpert. | immediately after asking the medical history and collecting the result of TB diagnosis
  According to the patients' health-seeking pathways, calculate the test coverage rates including anti fast bacteria smear, tuberculosis culture, and GeneXpert in different clinical institutions. The test coverage rates is acquired by recording the laboratory test reports in medical systems or paper version from patients.
The correlation between the use of fluoroquinolones as anti-infection treatment before tuberculosis diagnosis confirmed and the diagnosis delay of the pulmonary tuberculosis | immediately after asking the medical history and collecting the result of TB diagnosis
  We collect the fluoroquinolones use evidence of each patients in different clinical institutions by asking the past medical histories and reviewing paper reports from patients as well as medical system. Then use logistic correlation to find the relation between the fluoroquinolones use history and the diagnosis delay of the pulmonary tuberculosis.
The sociodemographic characteristics of patients with or without pulmonary tuberculosis diagnosis delay. | immediately after asking the medical history and collecting the result of TB diagnosis
  Calculating the distribution of patients' sociodemographic characteristics and correlation between results above and pulmonary tuberculosis diagnosis delay. Patients' sociodemographic characteristics includes: age, sex, marriage status, nation, occupation, education status, annual family income per capita, underlying disease such as diabetes, habits of smoking and habits of drinking alcohol.
The rates of onset symptoms and its correlation to diagnosis delayed of pulmonary tuberculosis diagnosis confirmed patients. | immediately after asking the medical history and collecting the result of TB diagnosis
  According to the past medical history of each pulmonary tuberculosis diagnosis confirmed patients, we collect their onset symptoms and calculate the rate respectively. Then use logistic correlation to find the relation between the onset symptoms and the diagnosis delay of the pulmonary tuberculosis.

CONTACTS AND LOCATIONS:
Overall Officials: Wenhong Zhang, PHD, Principal Investigator — Huashan Hospita
Locations (20):
- China (20):
  - Anhui Province Hospital, Hefei, Anhui
  - The Third People's Hospital of Shenzhen, Shenzhen, Guangdong
  - Beihai Tuberculosis Hospital, Beihai, Guangxi
  - Guiyang Public Health Clinical Center, Guiyang, Guizhou
  - The 2th Hospital of Daqing, Daqing, Hei Longjiang
  - Henan Province Infectious Diseases Hospital, Zhengzhou, Henan
  - Wuhan Medical Treatment Center, Wuhan, Hubei
  - The First People's Hospital of Huaihua, Huaihua, Hunan
  - The First People's Hospital of Taicang, Taicang, Jiangsu
  - Xuzhou Infectious Diseases Hospital Huimei Liu, Xuzhou, Jiangsu
  - Jiangxi Province Chest Hospital, Nanchang, Jiangxi
  - Changchun Infectious Diseases Hospital, Changchun, Jilin
  - Shandong Province Chest hospital, Jinan, Shandong
  - 905th Hospital of PLA Navy, Shanghai, Shanghai Municipality
  - Shanghai Public Health Clinical Center, Shanghai, Shanghai Municipality
  - Xian Chest Hospital, Xian, Shanxi
  - Southwest Medical University Affiliated Hospital, Luzhou, Sichuan
  - Qiubei People's Hospital, Jinping, Yunnan
  - Hangzhou Red Cross Hospital, Hangzhou, Zhejiang
  - Wenzhou Central Hospital, Wenzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes
We would like to share the study protocol and statistical analysis plan.
Supporting Information: Study Protocol, SAP
Time Frame: The data is available currently without expiry date.
Access Criteria: Please contact y_li11@fudan.edu.cn

REFERENCES:
- [Result] Liu R, Li J, Tan Y, Shang Y, Li Y, Su B, Shu W, Pang Y, Gao M, Ma L. Multicenter evaluation of the acid-fast bacillus smear, mycobacterial culture, Xpert MTB/RIF assay, and adenosine deaminase for the diagnosis of tuberculous peritonitis in China. Int J Infect Dis. 2020 Jan;90:119-124. doi: 10.1016/j.ijid.2019.10.036. Epub 2019 Nov 4. PMID 31693941
- [Result] Martinez L, Xu L, Chen C, Sekandi JN, Zhu Y, Zhang C, Whalen CC, Zhu L. Delays and Pathways to Final Tuberculosis Diagnosis in Patients from a Referral Hospital in Urban China. Am J Trop Med Hyg. 2017 May;96(5):1060-1065. doi: 10.4269/ajtmh.16-0358. Epub 2017 Feb 13. PMID 28193742
- [Result] Hogan CA, Puri L, Gore G, Pai M. Impact of fluoroquinolone treatment on delay of tuberculosis diagnosis: A systematic review and meta-analysis. J Clin Tuberc Other Mycobact Dis. 2016 Dec 13;6:1-7. doi: 10.1016/j.jctube.2016.12.001. eCollection 2017 Jan. PMID 31723692
- [Result] Storla DG, Yimer S, Bjune GA. A systematic review of delay in the diagnosis and treatment of tuberculosis. BMC Public Health. 2008 Jan 14;8:15. doi: 10.1186/1471-2458-8-15. PMID 18194573
- [Result] Hanson CL, Osberg M, Brown J, Durham G, Chin DP. Conducting Patient-Pathway Analysis to Inform Programming of Tuberculosis Services: Methods. J Infect Dis. 2017 Nov 6;216(suppl_7):S679-S685. doi: 10.1093/infdis/jix387. PMID 29117350
- [Result] Hanson C, Osberg M, Brown J, Durham G, Chin DP. Finding the Missing Patients With Tuberculosis: Lessons Learned From Patient-Pathway Analyses in 5 Countries. J Infect Dis. 2017 Nov 6;216(suppl_7):S686-S695. doi: 10.1093/infdis/jix388. PMID 29117351
- [Result] Farhat MR, Jacobson KR, Franke MF, Kaur D, Murray M, Mitnick CD. Fluoroquinolone Resistance Mutation Detection Is Equivalent to Culture-Based Drug Sensitivity Testing for Predicting Multidrug-Resistant Tuberculosis Treatment Outcome: A Retrospective Cohort Study. Clin Infect Dis. 2017 Oct 15;65(8):1364-1370. doi: 10.1093/cid/cix556. PMID 29017248
- [Result] Lewinsohn DM, Leonard MK, LoBue PA, Cohn DL, Daley CL, Desmond E, Keane J, Lewinsohn DA, Loeffler AM, Mazurek GH, O'Brien RJ, Pai M, Richeldi L, Salfinger M, Shinnick TM, Sterling TR, Warshauer DM, Woods GL. Official American Thoracic Society/Infectious Diseases Society of America/Centers for Disease Control and Prevention Clinical Practice Guidelines: Diagnosis of Tuberculosis in Adults and Children. Clin Infect Dis. 2017 Jan 15;64(2):111-115. doi: 10.1093/cid/ciw778. PMID 28052967
- [Result] GBD Tuberculosis Collaborators. Global, regional, and national burden of tuberculosis, 1990-2016: results from the Global Burden of Diseases, Injuries, and Risk Factors 2016 Study. Lancet Infect Dis. 2018 Dec;18(12):1329-1349. doi: 10.1016/S1473-3099(18)30625-X. PMID 30507459
- [Result] Mijiti P, Yuehua L, Feng X, Milligan PJ, Merle C, Gang W, Nianqiang L, Upur H. Prevalence of pulmonary tuberculosis in western China in 2010-11: a population-based, cross-sectional survey. Lancet Glob Health. 2016 Jul;4(7):e485-94. doi: 10.1016/S2214-109X(16)30074-2. Epub 2016 Jun 6. PMID 27283762